CLINICAL TRIAL: NCT04230720
Title: Impact of Lubrication With Artificial Tears on Biometry Measurements for Cataract Surgery
Brief Title: Effect of Artificial Tears on Biometry
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Stopped due to COVID-19.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-11021101
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Cataract
Keywords: biometry measurement; artificial tear; cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Artificial Tears (Experimental): One eye of each participant is randomized to receive Systane Complete artificial tears 4 times a day for 14 days
  Interventions: Drug: Systane Complete
- No Artificial Tears (No Intervention): One eye of each participant is randomized to receive no artificial tears for 14 days

INTERVENTIONS:
Drug: Systane Complete — 1 drop 4 times a day for 14 days
  Arms: Artificial Tears

SUMMARY:
The purpose of this study is to determine if measurements for cataract surgery are improved with use of additional lubrication with artificial tears. The research study is being done to optimize measurements and provide patients with the best visual outcomes after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Documentation of bilateral age-related senile cataracts diagnosis

Exclusion Criteria:

* Patients currently using regularly scheduled artificial tears. Patients with infrequent or irregular use of artificial tears may not be excluded from the study.
* Patients using contact lenses.
* Patients with any other surface pathology affecting corneal biometric measurements determined with slit-lamp examination or medical history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Baseline in Keratometry Values (K1 and K2) | Baseline, Day 14
  The change in keratometry (K) values (K1 and K2) in all subjects
Change in Baseline in Axis of Astigmatism | Baseline, Day 14
  The change in axis of astigmatism in all subjects

SECONDARY OUTCOMES:
Change in Baseline Calculated Intraocular Lens Power | Baseline, Day 14
  The change in intraocular lens power calculation in all subjects
Change in Keratometry Values (K1 and K2) in Ocular Surface Disease Subjects | Baseline, Day 14
  The change in keratometry (K) values (K1 and K2) in a subset of subjects that were positive for ocular surface disease on the American Society of Cataract and Refractive Surgery (ASCRS) modified Standardized Patient Evaluation of Eye Dryness (SPEED2) questionnaire
Change in Axis of Astigmatism in Ocular Surface Disease Subjects | Baseline, Day 14
  The change in axis of corneal astigmatism in a subset of subjects that were positive for ocular surface disease on the American Society of Cataract and Refractive Surgery (ASCRS) modified Standardized Patient Evaluation of Eye Dryness (SPEED2) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Brissette, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Ophthalmology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No